CLINICAL TRIAL: NCT02303678
Title: Phase I Single-Center, Dose Escalation Study of D2C7-IT Administered Intratumorally Via Convection-Enhanced Delivery for Adult Patients With Recurrent Malignant Glioma
Brief Title: D2C7 for Adult Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Darell Bigner (Other)
Responsible Party: Sponsor-Investigator, Darell Bigner, Edwin L. Jones, Jr. and Lucille Finch Jones Cancer Research Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053325
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Malignant Glioma; Brain Tumor, Recurrent
Keywords: D2C7; Randazzo; Bigner; Pro00053325; recurrent malignant glioma; Landi
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — D2C7-(scdsFv)-PE38KDEL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- D2C7-IT (Experimental): Recurrent malignant glioma patients will receive D2C7-IT, delivered intratumorally by CED following confirmatory diagnostic biopsy.
  Interventions: Drug: D2C7-IT

INTERVENTIONS:
Drug: D2C7-IT — D2C7-IT is a single-chain fragment variable (scFv) monoclonal antibody (Mab) fragment immunotoxin with high binding affinity for both EGFRwt- and EGFRvIII-expressing glioblastoma multiforme (GBM) cells.

SUMMARY:
This is a Phase I study to determine the maximum tolerated dose (MTD) and/or recommended phase II dose of D2C7-IT (D2C7 Immunotoxin) when delivered intratumorally by convection-enhanced delivery (CED) to recurrent World Health Organization (WHO) grade III and IV malignant glioma patients, and/or to determine what dose will be considered in a Phase II trial. Patients with recurrent WHO grade III and IV malignant glioma who meet eligibility criteria will be enrolled into the study. Immediately following the stereotactically-guided tumor biopsy conducted as standard of care, up to three additional core biopsies will be obtained for molecular genetic testing. After these biopsies are obtained, subjects will have up to 2 catheters inserted. If the biopsy indicates a proven diagnosis of recurrent malignant glioma (diagnosis results are typically received within 24-48 hours following biopsy), the investigators will proceed with the D2C7-IT infusion. If no tumor is identified, the catheters will be removed. A continuous intratumoral infusion of D2C7-IT will be administered over 72 hours while in the hospital.

DETAILED DESCRIPTION:
This is a Phase I study to determine the maximum tolerated dose (MTD) of D2C7-IT, when delivered intratumorally by convection-enhanced delivery (CED) following confirmatory diagnostic biopsy in recurrent World Health Organization (WHO) grade III and IV malignant glioma patients, and/or to determine what dose will be considered in a phase II trial. The patient will remain in the hospital during the entire infusion. At the completion of the infusion, the catheters will be removed within 6 hours and a CT scan will be obtained after the catheters are pulled. The patient will be observed in hospital for a minimum of another 6 hours.

A two-stage continual reassessment method (CRM) design will be used to determine the MTD of D2C7-IT where the first stage involves dose escalation in successive patients until an initial dose-limiting toxicity (DLT) is observed. Cohorts of 2 patients will be accrued to this study within both stages of the trial. The first patient of each cohort will be observed through the completion of the D2C7-IT infusion, before additional patients in that cohort are treated. Once the optimal dose level of D2C7-IT is determined (dose escalation completed), a total of 27 recurrent patients with WHO grade IV malignant glioma patients will be treated at that dose level as a dose expansion cohort.

Following D2C7-IT infusion, subjects will be evaluated in clinic at 2 weeks for adverse events and followed at 4 and 8 weeks and every 8 weeks thereafter until 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a recurrent supratentorial WHO grade III or IV malignant glioma based on imaging studies;
* Prior histopathology consistent with a supratentorial WHO grade III or IV malignant glioma;
* Following biopsy, prior to administration of D2C7-IT, the presence of recurrent tumor must be confirmed by histopathological analysis;
* Age ≥ 18 years of age;
* Karnofsky Performance Status (KPS) ≥ 70%;
* Laboratory Values:

  * Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion;
  * Hemoglobin ≥ 9 gm/dL prior to biopsy;
  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 prior to biopsy;
  * Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) prior to biopsy;
  * Liver Function: Total bilirubin ≤ 1.5 x ULN prior to biopsy (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.); AST (aspartate aminotransferase)/ALT (alanine aminotransferase) ≤ 2.5 x the ULN prior to biopsy;
  * Prothrombin (PT) and activated Partial Thromboplastin Time (aPTT) ≤ 1.2 x upper limit of normal (ULN) prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anti-coagulation will be held in the peri-operative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy;
* Ability to comply with study and follow-up procedures;

  * If the patient is a sexually active female of child bearing potential, whose partner is male, or if the patient is a sexually active male, whose partner is a female of child bearing potential, the patient must agree to use appropriate contraceptive measures for the duration of the treatment of the tumor and for 6 months afterwards as stated in the informed consent. Female patients of child bearing potential must have a negative serum pregnancy test at the time of screening and within 48 hours of starting the D2C7-IT infusion
* Patients will sign an IRB-approved informed consent form prior to any study-related procedures.
* Able to undergo brain MRI with and without contrast.

Exclusion Criteria:

* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin;
* Pregnant or breastfeeding;
* Patients with contrast-enhancing tumor component crossing the midline, actively growing multi-focal tumor, infratentorial tumor or extensive tumor dissemination (subependymal or leptomeningeal);
* Patients with clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment;
* Patients with a known severe allergy to Gadolinium-DTPA. Patients with mild allergies (e.g., rash only) will be pretreated with acetaminophen and diphenhydramine prior to injection of the contrast agent;
* Unstable systemic disease in the opinion of the treating physician, for example active infection requiring IV antibiotics;
* Patients on greater than 4mg per day of dexamethasone within the 2 weeks prior to admission for D2C7-IT infusion;
* Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups);
* Patients who have not completed standard of care treatment prior to participation in this trial, i.e. surgical procedure and radiation therapy (at least 59 Gy). Note: If tumor is unmethylated, patients are not mandated to have received chemotherapy prior to participation in this trial. However, if tumor is methylated, patients must have received at least one chemotherapy regimen prior to participation in this trial.
* Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation;
* Treated with immunotherapeutic agents within 4 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy;
* Treated with antiangiogenic agents (like bevacizumab) within 4 weeks before biopsy;
* Treated with alkylating agents within 4 weeks before enrollment (6 weeks for nitrosoureas) or treated within 1 week before enrollment with daily or metronomic chemotherapy, unless the patient has recovered from the expected toxic effects of such therapy;
* Prior chemotherapy (non-alkylating agents) within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and/or recommended phase II dose of D2C7-IT | 2 weeks after D2C7 administration
  The MTD is the dose that results in an estimated DLT rate based upon the CRM model that is nearest to the target DLT rate of 0.25. DLTs include any ≥ Gr.3 non-hematologic toxicities, any ≥ Gr.3 neurological toxicities, and any ≥ Gr.3 hematologic toxicities that do not resolve to pre-treatment baseline or ≤ Gr.1 within 2 weeks or any toxicity that resolves within the 2 week period, but then recurs during that same 2 week period. Adverse events will be collected using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  OS is defined at the time between administration of D2C7-IT and death. For patients alive, OS will be censored at the time of last follow-up. Kaplan-Meier methods will be used to estimate median OS and PFS.
Association between EGFRvIII and EGFRwt expression and PFS and OS. | 3 years
  Cox proportional hazards models will explore the relationship between EGFRvIII and EGFRwt expression as measured by immunohistochemistry (IHC), polymerase chain reactions (PCR), and fluorescence in situ hybridization (FISH) and PFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Landi, MD, Principal Investigator — Preston Robert Tisch Brain Tumor Center at Duke University Medical Center
Locations (1):
- Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

REFERENCES:
- [Derived] Bao X, Pastan I, Bigner DD, Chandramohan V. EGFR/EGFRvIII-targeted immunotoxin therapy for the treatment of glioblastomas via convection-enhanced delivery. Receptors Clin Investig. 2016;3(4):e1430. doi: 10.14800/rci.1430. PMID 28286803
- [Derived] Chandramohan V, Pegram CN, Piao H, Szafranski SE, Kuan CT, Pastan IH, Bigner DD. Production and quality control assessment of a GLP-grade immunotoxin, D2C7-(scdsFv)-PE38KDEL, for a phase I/II clinical trial. Appl Microbiol Biotechnol. 2017 Apr;101(7):2747-2766. doi: 10.1007/s00253-016-8063-x. Epub 2016 Dec 24. PMID 28013405
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/